CLINICAL TRIAL: NCT03753932
Title: Patients With Head and Neck Cancer Treated by Radiotherapy: The Impact of Fixed Dentures on Wellbeing and Oral Health Related Quality of Life
Brief Title: Impact of Fixed Dentures in Head and Neck Cancer (IMFDHAC)
Acronym: IMFDHAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Jönköping County (Other Government)
Collaborators: School of Health Sciences, Jönköping University, Jönköping Sweden (Unknown); Malmö University (Other)
Responsible Party: Principal Investigator, Carl-Otto Brahm, LDS, PhD, LDS, PhD, specialist in oral medicine, Region Jönköping County
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FORSS-385261; FORSS-341741 (Other Grant/Funding Number: FORSS); FUTURUM-265981 (Other Grant/Funding Number: Futurum)
Record Dates: First submitted 2018-11-07; First posted 2018-11-27 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2021-03

CONDITIONS: Head and Neck Neoplasms; Dental Prosthesis; Dentures; Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Single group for the control vs. intervention group. Crossover model within the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Dentures (fixed oral prosthesis) compared with standard treatment (removable oral prosthesis).
  Interventions: Device: Fixed prosthodontics

INTERVENTIONS:
Device: Fixed prosthodontics — The intervention takes place six months after finishing radiotherapy.

SUMMARY:
The purpose of the multi centre study is to evaluate an intervention, which means that patients undergoing radiotherapy for head and neck cancer will receive fixed dentures in accordance with the Public Health Care fee system with regard to well-being and oral health related quality of life.

Hypotheses: the intervention will improve oral health related quality of life, general wellbeing, and nutrition in patients treated by radiotherapy, with or without combination of chemotherapy or surgery against head and neck cancer.

DETAILED DESCRIPTION:
The oncological care is multidisciplinary. In the investigation phase for radiotherapy, the Ear-Nose-Throat (ENT) physician refer the patient for a dental examination. Any dental infections are treated to reduce the risk of radiation-related infections that may occur after cancer treatment. This may mean that infected but symptom-free teeth, which the patient experiences as healthy need to be removed. This prophylactic dental treatment is charged according to the Public Health Care fee system.

The study will take place in one major and in four middle sized counties in Sweden. The intervention will include 30 patients with head and neck cancer recruited from a Department of Maxillofacial and Oral Surgery (the City of Jönköping, Jönköping County Council), and from the Department of Orofacial Medicine (the City of Stockholm, Stockholm County Council). Another 30 patients with the same disease will be matched controls recruited from another Department of Maxillofacial and Oral Surgery (the City of Linköping, County Council of Östergötland) and from five Departments of Orofacial Medicine (the Cities of Kalmar, Oskarshamn, and Västervik, Kalmar County Council; the City of Växjö, Kronoberg County Council).

The project consists of three sub-studies: A quantitative study; a qualitative study; and a health economics study. About 30 patients will be included in the intervention group, as well as about 30 matched control patients. Data collection will take place with questionnaires (SF-36, EQ-5D, OHIP-14, GOHAI, JFLS-8, OAS) and interviews.

Patients recruited to the intervention group will be treated prosthodontically with removable and later with fixed dentures, thus acting as their own controls.

If possible but not necessary, those controls may be prosthodontically rehabilitated with temporary removable dentures.

The inclusion criteria are patients with head and neck tumours considered to receive radiotherapy, with or without combination of chemotherapy or surgery, good oncological prognosis at baseline. After referral from an ENT-specialist, those patients being diagnosed with dental infections and therapy planned for dental extraction(s) will be included.

The following general exclusion criteria will be applied: any communication problems; any comorbidity with poor prognosis; poor oncological prognosis at baseline; imminent risk of recurrence; any technical, biological, or any other reasonable obstacle of treating patients with fixed dentures; and finally patients in the matched control group financing fixed oral prosthesis themselves.

Background data like sex, age, diagnosis, TNM-classification, hyposalivation, vertical jaw mobility, dysphagia, number and sites of extracted teeth, and weight will be investigated.

Statistical analysis, quantitative and qualitative, will show differences in well-being and mouth-related quality of life between the different groups studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with head and neck tumours considered to receive radiotherapy, with or without combination of chemotherapy or surgery
* Good oncological prognosis at baseline.
* Patients diagnosed with dental infections and therapy planned for dental extraction(s).

Exclusion Criteria:

* Unwillingness to participate in the study.
* Patients with communication problems.
* Patients with comorbidity with poor prognosis.
* Patients with poor oncological prognosis at baseline.
* Patients with imminent risk of recurrence.
* Patients with any technical, biological, or any other reasonable obstacle of treating patients with fixed dentures
* Patients in the matched control group financing fixed oral prosthesis themselves.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Oral Health Related Quality of Life (OHRQL), OHIP-14, BL/T1 | Baseline
  Specific quality of life measured by the Oral Health Impact Profile (OHIP-14). OHRQL measurements are constructed to provide information about oral symptoms and related psychosocial and functional problems in dental public health perspectives as well as in clinical trials. Thus, when identifying and selecting a measure of OHRQL it is essential to use one with acceptable reliability and validity measuring the intended aims of the research. OHIP-14 is an instrument consisting of 14 items. Range 14 (better OHRQL) to 70 (worse OHRQL). It was designed to provide a comprehensive measure of the dysfunction, discomfort and disability attributed to oral conditions. Validated Swedish versions of the OHIP-14 are available.
Oral Health Related Quality of Life (OHRQL), OHIP-14, T2 | 6 months after completed radiotherapy
  Specific quality of life measured by the Oral Health Impact Profile (OHIP-14). OHRQL measurements are constructed to provide information about oral symptoms and related psychosocial and functional problems in dental public health perspectives as well as in clinical trials. Thus, when identifying and selecting a measure of OHRQL it is essential to use one with acceptable reliability and validity measuring the intended aims of the research. OHIP-14 is an instrument consisting of 14 items. Range 14 (better OHRQL) to 70 (worse OHRQL). It was designed to provide a comprehensive measure of the dysfunction, discomfort and disability attributed to oral conditions. Validated Swedish versions of the OHIP-14 are available.
Oral Health Related Quality of Life (OHRQL), OHIP-14, T3 | 12 months after completed radiotherapy
  Specific quality of life measured by the Oral Health Impact Profile (OHIP-14). OHRQL measurements are constructed to provide information about oral symptoms and related psychosocial and functional problems in dental public health perspectives as well as in clinical trials. Thus, when identifying and selecting a measure of OHRQL it is essential to use one with acceptable reliability and validity measuring the intended aims of the research. OHIP-14 is an instrument consisting of 14 items. Range 14 (better OHRQL) to 70 (worse OHRQL). It was designed to provide a comprehensive measure of the dysfunction, discomfort and disability attributed to oral conditions. Validated Swedish versions of the OHIP-14 are available.
Oral Health Related Quality of Life (OHRQL), GOHAI, BL/T1 | Baseline
  Specific quality of life measured by the General Oral Health Assessment Index (GOHAI) which is a 12-item instrument originally developed for use with older adult populations, although more recently it has been used with populations of younger adults. Range 12 (worse OHRQL) to 60 (better OHRQL). It measures oral functional problems and also assesses the psychosocial impacts associated with oral disease. A Swedish version has been validated.
Oral Health Related Quality of Life (OHRQL), GOHAI, T2 | 6 months after completed radiotherapy
  Specific quality of life measured by the General Oral Health Assessment Index (GOHAI) which is a 12-item instrument originally developed for use with older adult populations, although more recently it has been used with populations of younger adults. Range 12 (worse OHRQL) to 60 (better OHRQL). It measures oral functional problems and also assesses the psychosocial impacts associated with oral disease. A Swedish version has been validated.
Oral Health Related Quality of Life (OHRQL), GOHAI, T3 | 12 months after completed radiotherapy
  Specific quality of life measured by the General Oral Health Assessment Index (GOHAI) which is a 12-item instrument originally developed for use with older adult populations, although more recently it has been used with populations of younger adults. Range 12 (worse OHRQL) to 60 (better OHRQL). It measures oral functional problems and also assesses the psychosocial impacts associated with oral disease. A Swedish version has been validated.

SECONDARY OUTCOMES:
Wellbeing, Quality of Life (QoL), SF-36v2, BL/T1 | Baseline
  General quality of life measured by the SF-36 v2. SF-36v2 is a well established psychometric instrument with 36 items measuring eight domains of health-related quality of life: Physical function, physical role function, bodily pain, general health, vitality, social function, emotional role function, mental health. The two comprehensive indices - physical health and mental health - can be estimated for. Range 0 (worse QoL) to 100 (better QoL). The instrument is translated and validated into Swedish.
Wellbeing, Quality of Life (QoL), SF-36v2, T2 | 6 months after completed radiotherapy
  General quality of life measured by the SF-36 v2. SF-36v2 is a well established psychometric instrument with 36 items measuring eight domains of health-related quality of life: Physical function, physical role function, bodily pain, general health, vitality, social function, emotional role function, mental health. The two comprehensive indices - physical health and mental health - can be estimated for. Range 0 (worse QoL) to 100 (better QoL). The instrument is translated and validated into Swedish.
Wellbeing, Quality of Life (QoL), SF-36v2, T3 | 12 months after completed radiotherapy
  General quality of life measured by the SF-36 v2. SF-36v2 is a well established psychometric instrument with 36 items measuring eight domains of health-related quality of life: Physical function, physical role function, bodily pain, general health, vitality, social function, emotional role function, mental health. The two comprehensive indices - physical health and mental health - can be estimated for. Range 0 (worse QoL) to 100 (better QoL). The instrument is translated and validated into Swedish.
Wellbeing, Health Related Quality of Life (HRQoL), EQ-5D, BL/T1 | Baseline
  General quality of life measured by the EQ-5D which is an instrument containing five items measuring mobility, self-care, pain, role function, and anxiety/depression. There is also one item considering change of health condition and a VAS scale for general health. There is no total score, however there are different levels of HRQoL: Level 1. better HRQoL; Level 3. worse HRQoL. This instrument is translated and validated into Swedish.
Wellbeing, Health Related Quality of Life (HRQoL), EQ-5D, T2 | 6 months after completed radiotherapy
  General quality of life measured by the EQ-5D which is an instrument containing five items measuring mobility, self-care, pain, role function, and anxiety/depression. There is also one item considering change of health condition and a VAS scale for general health. There is no total score, however there are different levels of HRQoL: Level 1. better HRQoL; Level 3. worse HRQoL. This instrument is translated and validated into Swedish.
Wellbeing, Health Related Quality of Life (HRQoL), EQ-5D, T3 | 12 months after completed radiotherapy
  General quality of life measured by the EQ-5D which is an instrument containing five items measuring mobility, self-care, pain, role function, and anxiety/depression. There is also one item considering change of health condition and a VAS scale for general health. There is no total score, however there are different levels of HRQoL: Level 1. better HRQoL; Level 3. worse HRQoL. This instrument is translated and validated into Swedish.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Malm, Assoc Prof, Study Director — School of Health and Science, Jönköping Sweden
Locations (1):
- Public Dental Health, Jönköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korfage A, Schoen PJ, Raghoebar GM, Roodenburg JL, Vissink A, Reintsema H. Benefits of dental implants installed during ablative tumour surgery in oral cancer patients: a prospective 5-year clinical trial. Clin Oral Implants Res. 2010 Sep;21(9):971-9. doi: 10.1111/j.1600-0501.2010.01930.x. PMID 20701621
- [Background] Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. Qual Health Res. 2005 Nov;15(9):1277-88. doi: 10.1177/1049732305276687. PMID 16204405
- [Result] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Result] Vissink A, Jansma J, Spijkervet FK, Burlage FR, Coppes RP. Oral sequelae of head and neck radiotherapy. Crit Rev Oral Biol Med. 2003;14(3):199-212. doi: 10.1177/154411130301400305. PMID 12799323
- [Result] Kielbassa AM, Hinkelbein W, Hellwig E, Meyer-Luckel H. Radiation-related damage to dentition. Lancet Oncol. 2006 Apr;7(4):326-35. doi: 10.1016/S1470-2045(06)70658-1. PMID 16574548
- [Result] Jham BC, da Silva Freire AR. Oral complications of radiotherapy in the head and neck. Braz J Otorhinolaryngol. 2006 Sep-Oct;72(5):704-8. doi: 10.1016/s1808-8694(15)31029-6. PMID 17221065
- [Result] Store G, Granstrom G. Osteoradionecrosis of the mandible: a microradiographic study of cortical bone. Scand J Plast Reconstr Surg Hand Surg. 1999 Sep;33(3):307-14. doi: 10.1080/02844319950159280. PMID 10505444
- [Result] Korfage A, Schoen PJ, Raghoebar GM, Bouma J, Burlage FR, Roodenburg JL, Vissink A, Reintsema H. Five-year follow-up of oral functioning and quality of life in patients with oral cancer with implant-retained mandibular overdentures. Head Neck. 2011 Jun;33(6):831-9. doi: 10.1002/hed.21544. Epub 2010 Dec 9. PMID 21560179
- [Result] Jager-Wittenaar H, Dijkstra PU, Vissink A, van der Laan BF, van Oort RP, Roodenburg JL. Malnutrition and quality of life in patients treated for oral or oropharyngeal cancer. Head Neck. 2011 Apr;33(4):490-6. doi: 10.1002/hed.21473. Epub 2010 Sep 7. PMID 20824806
- [Result] Dwivedi RC, Kazi RA, Agrawal N, Nutting CM, Clarke PM, Kerawala CJ, Rhys-Evans PH, Harrington KJ. Evaluation of speech outcomes following treatment of oral and oropharyngeal cancers. Cancer Treat Rev. 2009 Aug;35(5):417-24. doi: 10.1016/j.ctrv.2009.04.013. Epub 2009 May 29. PMID 19481871
- [Result] John MT, Slade GD, Szentpetery A, Setz JM. Oral health-related quality of life in patients treated with fixed, removable, and complete dentures 1 month and 6 to 12 months after treatment. Int J Prosthodont. 2004 Sep-Oct;17(5):503-11. PMID 15543905
- [Result] Lekholm U, Grondahl K, Jemt T. Outcome of oral implant treatment in partially edentulous jaws followed 20 years in clinical function. Clin Implant Dent Relat Res. 2006;8(4):178-86. doi: 10.1111/j.1708-8208.2006.00019.x. PMID 17100743
- [Result] Jemt T, Johansson J. Implant treatment in the edentulous maxillae: a 15-year follow-up study on 76 consecutive patients provided with fixed prostheses. Clin Implant Dent Relat Res. 2006;8(2):61-9. doi: 10.1111/j.1708-8208.2006.00003.x. PMID 16774591
- [Result] Andersson G, Andreasson L, Bjelkengren G. Oral implant rehabilitation in irradiated patients without adjunctive hyperbaric oxygen. Int J Oral Maxillofac Implants. 1998 Sep-Oct;13(5):647-54. PMID 9796148
- [Result] Shaw RJ, Sutton AF, Cawood JI, Howell RA, Lowe D, Brown JS, Rogers SN, Vaughan ED. Oral rehabilitation after treatment for head and neck malignancy. Head Neck. 2005 Jun;27(6):459-70. doi: 10.1002/hed.20176. PMID 15880417
- [Result] Sullivan M, Karlsson J, Ware JE Jr. The Swedish SF-36 Health Survey--I. Evaluation of data quality, scaling assumptions, reliability and construct validity across general populations in Sweden. Soc Sci Med. 1995 Nov;41(10):1349-58. doi: 10.1016/0277-9536(95)00125-q. PMID 8560302
- [Result] Persson LO, Karlsson J, Bengtsson C, Steen B, Sullivan M. The Swedish SF-36 Health Survey II. Evaluation of clinical validity: results from population studies of elderly and women in Gothenborg. J Clin Epidemiol. 1998 Nov;51(11):1095-103. doi: 10.1016/s0895-4356(98)00101-2. PMID 9817127
- [Result] Sullivan M, Karlsson J. The Swedish SF-36 Health Survey III. Evaluation of criterion-based validity: results from normative population. J Clin Epidemiol. 1998 Nov;51(11):1105-13. doi: 10.1016/s0895-4356(98)00102-4. PMID 9817128
- [Result] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Result] Larsson B, Johannesson A, Andersson IH, Atroshi I. The Locomotor Capabilities Index; validity and reliability of the Swedish version in adults with lower limb amputation. Health Qual Life Outcomes. 2009 May 23;7:44. doi: 10.1186/1477-7525-7-44. PMID 19463185
- [Result] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Result] Hagglin C, Berggren U, Hakeberg M, Edvardsson A, Eriksson M. Evaluation of a Swedish version of the OHIP-14 among patients in general and specialist dental care. Swed Dent J. 2007;31(2):91-101. PMID 17695054
- [Result] Larsson P, List T, Lundstrom I, Marcusson A, Ohrbach R. Reliability and validity of a Swedish version of the Oral Health Impact Profile (OHIP-S). Acta Odontol Scand. 2004 Jun;62(3):147-52. doi: 10.1080/00016350410001496. PMID 15370634
- [Result] Atchison KA, Dolan TA. Development of the Geriatric Oral Health Assessment Index. J Dent Educ. 1990 Nov;54(11):680-7. PMID 2229624
- [Result] Hagglin C, Berggren U, Lundgren J. A Swedish version of the GOHAI index. Psychometric properties and validation. Swed Dent J. 2005;29(3):113-24. PMID 16255355
- [Result] Larsson P. Methodological studies of orofacial aesthetics, orofacial function and oral health-related quality of life. Swed Dent J Suppl. 2010;(204):11-98. PMID 20623943
- [Result] Ohrbach R, Larsson P, List T. The jaw functional limitation scale: development, reliability, and validity of 8-item and 20-item versions. J Orofac Pain. 2008 Summer;22(3):219-30. PMID 18780535
- [Result] Larsson P, John MT, Nilner K, List T. Reliability and validity of the Orofacial Esthetic Scale in prosthodontic patients. Int J Prosthodont. 2010 May-Jun;23(3):257-62. PMID 20552093
- [Result] Larsson P, John MT, Nilner K, Bondemark L, List T. Development of an Orofacial Esthetic Scale in prosthodontic patients. Int J Prosthodont. 2010 May-Jun;23(3):249-56. PMID 20552092
- [Result] Gellrich NC, Schramm A, Bockmann R, Kugler J. Follow-up in patients with oral cancer. J Oral Maxillofac Surg. 2002 Apr;60(4):380-6; discussion 387-8. doi: 10.1053/joms.2002.31224. PMID 11928093

DOCUMENTS (1):
  • Study Protocol (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT03753932/Prot_000.pdf